CLINICAL TRIAL: NCT06135662
Title: Tunnel Technique Versus Coronally Advanced Flap Combined With a Connective Tissue Graft for the Treatment of Mandibular Gingival Recessions: A Randomized Clinical Trial
Brief Title: Comparing Tunnel Technique and CAF With CTG in Mandibular Gingival Recession Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Clinical Head Staff, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2023-01
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Gingival Recession Localized Moderate
Keywords: RT1; RT2; CAF; Tunnel Technique; Connective Tissue Graft; Gingival Recessions; CTG
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF + CTG (Active Comparator): This arm involves patients treated with the Coronally Advanced Flap (CAF) technique, a recognized method for treating gingival recession. As an active comparator, this arm serves to compare the effectiveness and outcomes of CAF against the alternative surgical method used in the study.
  Interventions: Procedure: CAF + CTG
- Tunnel Technique + CTG (Active Comparator): Patients in this arm receive the Tunnel Technique (TT) with Connective Tissue Grafts (CTG). Also an established method for gingival recession treatment, this arm acts as an active comparator to assess and compare the effectiveness of TT+CTG against the CAF technique.
  Interventions: Procedure: Tunnel Technique + CTG

INTERVENTIONS:
Procedure: CAF + CTG — Surgical techniques for mandibular gingival recession: coronally advanced flap + connective tissue graft. Participants undergo initial evaluations, including periodontal exams and digital imaging, followed by standardized pre-operative preparations. Post-surgery, uniform care includes pain management and oral hygiene instructions, with follow-ups to monitor healing and assess outcomes. Primary and secondary outcomes, like root coverage and patient-reported satisfaction, are consistently measured across groups. Standardized data collection and analysis procedures ensure reliable, comparable results, facilitating an effective comparison of the surgical methods' efficacy.
  Arms: CAF + CTG
Procedure: Tunnel Technique + CTG — Surgical techniques for mandibular gingival recession: tunnel technique + connective tissue graft. Participants undergo initial evaluations, including periodontal exams and digital imaging, followed by standardized pre-operative preparations. Post-surgery, uniform care includes pain management and oral hygiene instructions, with follow-ups to monitor healing and assess outcomes. Primary and secondary outcomes, like root coverage and patient-reported satisfaction, are consistently measured across groups. Standardized data collection and analysis procedures ensure reliable, comparable results, facilitating an effective comparison of the surgical methods' efficacy.
  Arms: Tunnel Technique + CTG

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of two different surgical techniques, the Coronally Advanced Flap (CAF) and the Tunnel Technique (TT) with Connective Tissue Grafts (CTG), in treating mandibular gingival recession. This study, focusing on healthy patients with RT1 and RT2 gingival recessions, aims to determine which surgical approach offers better root coverage for mandibular recession defects. Additionally, it seeks to understand the effects of these techniques on aspects such as keratinized tissue gain, vestibular depth, gingival thickness, and patient-reported outcomes. Participants in this trial will undergo one of the two surgical procedures and are expected to attend a total of six assessment visits. Researchers will compare the results from both groups, those treated with CAF and those with TT+CTG, to discern if one method is superior in achieving more effective root coverage, enhanced aesthetic appearance, and reduced discomfort associated with gingival recession.

DETAILED DESCRIPTION:
This clinical trial is designed to rigorously assess the effectiveness of two surgical techniques, the Coronally Advanced Flap (CAF) and the Tunnel Technique (TT) with Connective Tissue Grafts (CTG), in the treatment of mandibular gingival recession, specifically targeting RT1 and RT2 types of recessions. The primary objective of this study is to determine which of these approaches provides superior root coverage in managing mandibular recession defects. The secondary objectives include evaluating the impact of these treatments on keratinized tissue gain, changes in vestibular depth, variations in gingival thickness, and patient-reported outcomes such as pain and aesthetic satisfaction.

Healthy participants diagnosed with mandibular gingival recession will be enrolled and randomly assigned to undergo either the CAF or TT+CTG surgical procedure. The study will follow a structured timeline with a total of six assessment visits for each participant, scheduled at key intervals: 1 week, 2 weeks, 6 weeks, 3 months, and 6 months post-operation. These time points are chosen to effectively monitor both the immediate and the long-term results of the treatments.

The primary outcome measure, Mean Root Coverage (MRC), will be evaluated at each follow-up visit to quantify the extent of root coverage achieved by the respective surgical techniques. Secondary outcome measures include the assessment of Vestibular Depth (VD), Complete Root Coverage (CRC), changes in Keratinized Tissue Width (KT), and changes in Gingival Thickness (GT). These measures will provide a comprehensive understanding of the physiological and aesthetic impacts of the surgical interventions.

By comparing the outcomes from both treatment groups, the study aims to provide clear evidence on the effectiveness of CAF versus TT+CTG in treating mandibular gingival recession, guiding future clinical decisions and patient care strategies in periodontology.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years; periodontally and systemically healthy
* presence of RT1 and RT2 gingival recession defects
* recession in the mandibular arch
* recession ≥ 2mm in depth at the buccal aspect
* full-mouth plaque and bleeding score ≤ 20%
* no previous periodontal surgery
* presence of identifiable cemento-enamel junction (CEJ) (a step ≤1mm at the CEJ and/or presence of root abrasion, but with identifiable CEJ, will be accepted).

Exclusion Criteria:

* smokers ≥10 cigarettes a day
* contraindications for periodontal surgery
* medications known to affect the gingiva or interfere with wound healing
* pregnancy
* active orthodontic therapy
* caries or restorations in the area to be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Mean Root Coverage (MRC) | At 1 week, 2 weeks, 6 weeks, 3 months, and 6 months post-operation
  he Mean Root Coverage measures the percentage of exposed tooth root that has been covered by gum tissue after surgery, compared to before the treatment.

SECONDARY OUTCOMES:
Vestibular depth (VD) | At 1 week, 2 weeks, 6 weeks, 3 months, and 6 months post-operation
  Measurement of the depth of the vestibular area (the space between the inside of the lip/cheek and the gum) to assess changes post-surgery.
Complete Root Coverage (CRC) | At 1 week, 2 weeks, 6 weeks, 3 months, and 6 months post-operation
  Assessment of whether the entire exposed root surface is covered by gum tissue post-treatment.
change in Keratinized Tissue Width (KT) | At 1 week, 2 weeks, 6 weeks, 3 months, and 6 months post-operation
  Measurement of the width of keratinized tissue (gum tissue that is firmly attached to the bone) to note any changes following the surgical procedure.
change in gingival thickness (GT) | At 1 week, 2 weeks, 6 weeks, 3 months, and 6 months post-operation
  Assessment of the thickness of the gum tissue to evaluate changes after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Blasi, DDS MS, Principal Investigator — UIC Barcelona
Locations (1):
- UIC Barcelona - Clinica Universitaria de Odontologia, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchelli G, De Sanctis M. Treatment of multiple recession-type defects in patients with esthetic demands. J Periodontol. 2000 Sep;71(9):1506-14. doi: 10.1902/jop.2000.71.9.1506. PMID 11022782
- [Result] Cairo F, Nieri M, Cattabriga M, Cortellini P, De Paoli S, De Sanctis M, Fonzar A, Francetti L, Merli M, Rasperini G, Silvestri M, Trombelli L, Zucchelli G, Pini-Prato GP. Root coverage esthetic score after treatment of gingival recession: an interrater agreement multicenter study. J Periodontol. 2010 Dec;81(12):1752-8. doi: 10.1902/jop.2010.100278. Epub 2010 Jul 14. PMID 20629546